CLINICAL TRIAL: NCT00519857
Title: A Multinational, Multicenter, Randomized, Double-Blind, Parallel Group,Placebo Controlled Clinical Trial of the Effects of Tibolone (Org OD-14 1.25mg) on the Incidence of New Vertebral Fractures in Osteoporotic Postmenopausal Women.
Brief Title: Trial to Evaluate Tibolone in the Treatment of Osteoporosis (P06468)
Acronym: LIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P06468; 32962
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Tibolone
  Interventions: Drug: Tibolone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tibolone — 1.25 mg p.o, once daily for 3 years
  Other Names: OD-14
  Arms: 1
Drug: Placebo — Tablet p.o, once daily for 3 years
  Arms: 2

SUMMARY:
Tibolone 1.25 mg is an effective treatment for the prevention of osteoporosis and is expected to be effective in preventing fractures in osteoporotic women. Tibolone could be more acceptable for long-term use, in particular since it does not induce a regular withdrawal bleed.

The objective of this trial is to compare placebo and tibolone, a steroid with tissue specific activity, in the prevention of spinal fractures in women meeting the WHO criteria for osteoporosis or who have asymptomatic vertebral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent, and who were willing and able to make reasonable efforts to observe all clinical trial requirements were to be enrolled
* Subjects were to be postmenopausal (naturally or surgically) women, from 60 to 85 years of age (inclusive) at entry
* Screening BMD of the total hip and/or spine had to be equal to or lower than 2.5 SD T-score for subjects without an asymptomatic fracture or equal to or lower than -2.0 SD T-score for subjects with an asymptomatic fracture
* Subjects were to have a Body Mass Index (BMI) = 34 kg/m^2.

Exclusion Criteria:

Subjects with any of the following conditions were not to be enrolled into the trial:

* Recent acute vertebral fracture (diagnosed within the last year) documented by spinal radiograph requiring medication for osteoporosis treatment, in the judgment of the investigator
* More than two prevalent asymptomatic vertebral fractures at baseline
* Screening BMD of the total hip or spine lower than -4 SD T-score
* Unsuitable anatomy on spinal radiographs (lumbar and thoracic vertebrae) e.g., excessive scoliosis
* Not ambulatory
* History or presence of any malignancy within the past five years except for nonmelanoma skin cancer. Subjects with ever history of ovarian cancer or estrogen dependent tumors particularly breast or endometrial cancer were to be excluded
* Trans vaginal ultrasound (TVUS) endometrial double wall thickness >4 mm
* Unexplained abnormal vaginal bleeding in the past year prior to screening
* Abnormal cervical Papanicolaou (Pap) smear (including low grade squamous intraepithelial lesion (LSIL), high grade squamous intraepithelial lesion (HSIL), atypical squamous cells of undetermined significance (ASCUS), atypical glands of undetermined significance (AGCUS))
* Mammography finding that was suspicious of malignancy
* Bone disease other than osteoporosis such as Paget's disease, osteomalacia, hyperparathyroidism, or bone metastases
* Treatment with anabolic steroids, calcitonin, raloxifene, tamoxifen, or calcitriol within the last six months prior to screening BMD or spinal X-ray measurements.
* Treatment with systemic estrogen and/or progestin within the last three months prior to screening BMD or spinal X-ray measurements (occasional use of estriol containing vaginal cream was allowed)
* Treatment with bisphosphonates for one month or more within the last year
* Ever use of estrogen and/or progestin containing implants

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4534 (Actual)
Dates: Start 2001-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter was reduction in incident new vertebral fractures assessed by spinal radiographs (anterior-posterior and lateral) | 3 years

SECONDARY OUTCOMES:
Bone mineral density of lumbar vertebrae (L1-L4) and left proximal femur for total hip density measured by means of dual-energy X-ray absorptiometry (DXA). | 3 years

REFERENCES:
- [Derived] Cummings SR, Ettinger B, Delmas PD, Kenemans P, Stathopoulos V, Verweij P, Mol-Arts M, Kloosterboer L, Mosca L, Christiansen C, Bilezikian J, Kerzberg EM, Johnson S, Zanchetta J, Grobbee DE, Seifert W, Eastell R; LIFT Trial Investigators. The effects of tibolone in older postmenopausal women. N Engl J Med. 2008 Aug 14;359(7):697-708. doi: 10.1056/NEJMoa0800743. PMID 18703472